CLINICAL TRIAL: NCT00368277
Title: A 36 Week Randomized, Double-blind, Parallel Group, Multi-center, Active-controlled, Optional Titration Study Comparing an Aliskiren-based Regimen to a Ramipril-based Regimen in Patients ≥ 65 Years Old With Systolic Essential Hypertension
Brief Title: A Safety and Efficacy Trial of Aliskiren 150mg , 300 mg Compared to Ramipril 5mg, 10mg in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2344
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Results first posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-02

CONDITIONS: Hypertension
Keywords: Systolic hypertension; hypertension; aliskiren; blood pressure; ramipril; HTN
MeSH Terms: conditions — Hypertension; Isolated Systolic Hypertension | interventions — aliskiren; Ramipril; Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aliskiren-based regimen (Experimental): Aliskiren 150 mg; aliskiren 300 mg; aliskiren 300mg + hydrochlorothiazide 12.5 mg; aliskiren 300 mg + hydrochlorothiazide 25 mg; aliskiren 300 mg + hydrochlorothiazide 25 mg + amlodipine 5 mg; aliskiren 300 mg + hydrochlorothiazide 25 mg + amlodipine 10 mg
  Interventions: Drug: Aliskiren; Drug: Hydrochlorothiazide; Drug: Amlodipine
- Ramipril-based regimen (Active Comparator): Ramipril 5 mg; Ramipril 10 mg; Ramipril 10 mg + hydrochlorothiazide 12.5 mg; Ramipril 10 mg + hydrochlorothiazide 25 mg; Ramipril 10 mg + hydrochlorothiazide 25 mg + amlodipine 5 mg; Ramipril 10 mg + hydrochlorothiazide 25 mg + amlodipine 10mg
  Interventions: Drug: Ramipril; Drug: Hydrochlorothiazide; Drug: Amlodipine

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 150 mg and 300 mg tablets taken orally, once a day in the morning
  Arms: Aliskiren-based regimen
Drug: Ramipril — Ramipril 5 mg and 10 mg capsules taken orally, once a day in the morning
  Arms: Ramipril-based regimen
Drug: Hydrochlorothiazide — Hydrochlorothiazide 12.5 or 25 mg capsules taken orally, once a day in the morning
Drug: Amlodipine — Amlodipine 5 mg or 10 mg tablets taken orally, once a day in the morning

SUMMARY:
Evaluate the systolic blood pressure lowering effect of aliskiren 150mg and 300mg compared to ramipril 5mg and 10mg in elderly patients with essential systolic hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients ≥ 65 years old.
* Patients with essential hypertension with an msSBP ≥ 140 mmHg and < 180 mmHg, and msDBP < 110 mmHg at Visits 2 and 3. (Visit 201 was deleted by the Administrative Changes document.)
* Patients must have had a difference in msSBP of ≤ 20 mmHg between Visit 3 and the visit immediately prior to Visit 3.
* Patients who were eligible and able to participate in the study, and who consented to do so after the purpose and nature of the investigation had been explained to them (written informed consent).

Exclusion Criteria:

* History of renal artery stenosis.
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* History of hypertensive encephalopathy.
* Current diagnosis of heart failure (New York Heart Association Class III-IV).
* History of transient ischemic cerebral attack or cerebrovascular accident within 6 months.
* History of myocardial infarction, bypass surgery, or any percutaneous coronary intervention within 6 months.
* Current unstable angina pectoris. Patients on a stable dose of oral or topical nitrates or beta blockers for angina were acceptable.
* Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia.
* Clinically significant valvular heart disease.
* Concurrent use of any antihypersensitive medications except a stable dose 3 months prior to visit 1 of alpha adrenergic blockers for benign prostatic hypertrophy (e.g., Flomax for BPH), beta blockers for angina, or beta blockers ophthalmic preparations.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 901 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Wang GM, Li LJ, Tang WL, Wright JM. Renin inhibitors versus angiotensin converting enzyme (ACE) inhibitors for primary hypertension. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD012569. doi: 10.1002/14651858.CD012569.pub2. PMID 33089502

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren Based Treatment Regimen: Aliskiren 150 mg; aliskiren 300 mg; aliskiren 300mg + hydrochlorothiazide 12.5 mg; aliskiren 300 mg + hydrochlorothiazide 25 mg; aliskiren 300 mg + hydrochlorothiazide 25 mg + amlodipine 5 mg; aliskiren 300 mg + hydrochlorothiazide 25 mg + amlodipine 10 mg
- Ramipril Based Treatment Regimen: Ramipril 5 mg; Ramipril 10 mg; Ramipril 10 mg + hydrochlorothiazide 12.5 mg; Ramipril 10 mg + hydrochlorothiazide 25 mg; Ramipril 10 mg + hydrochlorothiazide 25 mg + amlodipine 5 mg; Ramipril 10 mg + hydrochlorothiazide 25 mg + amlodipine 10mg
Period: Overall Study
Arm/Group | Aliskiren Based Treatment Regimen | Ramipril Based Treatment Regimen
Started | 457 | 444
Completed | 344 | 336
Not Completed | 113 | 108
Not completed — Adverse Event | 33 | 49
Not completed — Death | 2 | 1
Not completed — Unsatisfactory therapeutic effect | 31 | 24
Not completed — Protocol deviation | 7 | 0
Not completed — Patient withdrew consent | 32 | 28
Not completed — Lost to Follow-up | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren Based Treatment Regimen | Ramipril Based Treatment Regimen | Total
Number analyzed (Participants) | 457 | 444 | 901
Age Continuous [Mean (Standard Deviation); unit: years] | 72.0 (5.56) | 72.2 (5.62) | 72.1 (5.58)
Age, Customized [Number; unit: participants]
  65 - 74 years | 312 | 296 | 608
  75 years and older | 145 | 148 | 293
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 235 | 237 | 472
  Male | 222 | 207 | 429

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure to Week 12
Time Frame: Baseline and Week 12
Population: Intent to treat (ITT), Last Observation Carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren Based Treatment Regimen | Ramipril Based Treatment Regimen
Number analyzed (Participants) | 451 | 439
mm Hg | -13.96 (0.754) [-15.15 to -12.13] | -11.64 (0.759) [-12.76 to -9.90]

2. Secondary Outcome: Percentage of Patients With Cough
Time Frame: Weeks 12 and 36
Population: Safety population
Measure: Number; unit: Percentage of Participants
Arm/Group | Aliskiren Based Treatment Regimen | Ramipril Based Treatment Regimen
Number analyzed (Participants) | 452 | 444
Percentage of Participants
  Week 12 | 3.1 (0.788) | 9.9 (0.794)
  Week 36 | 4.4 | 14.2

3. Secondary Outcome: Percentage of Patients Achieving Blood Pressure Control at Weeks 12 and 36 Endpoints
Description: Blood pressure control is defined as a mean sitting blood pressure < 140/90 mm Hg
Time Frame: Weeks 12 and 36
Population: intent to treat (ITT), last observation carried forward (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren Based Treatment Regimen | Ramipril Based Treatment Regimen
Number analyzed (Participants) | 451 | 440
Percentage of participants
  week 12 endpoint | 46.3 | 39.3
  week 36 endpoint | 65.6 | 57.5

4. Secondary Outcome: Change From Baseline in the Mean Sitting Diastolic Blood Pressure to Week 36
Time Frame: Baseline and week 36
Population: Intent to treat (ITT), Last Observation Carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren Based Treatment Regimen | Ramipril Based Treatment Regimen
Number analyzed (Participants) | 451 | 439
mm Hg | -8.24 (0.409) | -7.02 (0.411)

ADVERSE EVENTS:
Time Frame: 36 weeks
Groups:
- Aliskiren: Aliskiren based regimen
- Ramipril: Ramipril based regimen
Arm/Group | Aliskiren | Ramipril
Serious Adverse Events (participants affected / at risk) | 35/452 | 27/444
Other Adverse Events (participants affected / at risk) | 170/452 | 181/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=452) | Ramipril (N=444)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Trifascicular block (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Thyroid mass (Endocrine disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Eye movement disorder (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Aphagia (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 3
Oedema peripheral (General disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Myringitis bullous (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anoxic encephalopathy (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 4
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren (N=452) | Ramipril (N=444)
Diarrhoea (Gastrointestinal disorders) | 29 | 22
Fatigue (General disorders) | 28 | 20
Nasopharyngitis (Infections and infestations) | 23 | 20
Upper respiratory tract infection (Infections and infestations) | 35 | 28
Urinary tract infection (Infections and infestations) | 17 | 24
Dizziness (Nervous system disorders) | 34 | 37
Headache (Nervous system disorders) | 42 | 40
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.